CLINICAL TRIAL: NCT05570045
Title: Study the Efficiency of Oral Nutritional Supplementation on Anthropometric Indicators, Nutrition Status, Digestive Disorders, Anorexic and Upper Respiratory Infections in Children
Brief Title: Improvement of Nutrition Status, Digestive Conditions, and Upper Respiratory Infections by Using Oral Nutritional Supplementation on Children in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tu Nguyen Song (Other Government)
Responsible Party: Sponsor-Investigator, Tu Nguyen Song, Head of Division Planning, National Institute of Nutrition, Vietnam
Organization: National Institute of Nutrition, Vietnam (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: COLOS-NIN
Record Dates: First submitted 2022-09-26; First posted 2022-10-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Wasting; Undernutrition; Malnourished; Malnutrition
Keywords: children; oral nutrition supplementation; anorexic; anorexia nervosa; digestive disorders; upper respiratory infections; nutrition status; wasting
MeSH Terms: conditions — Cachexia; Malnutrition; Anorexia; Anorexia Nervosa; Digestive System Diseases; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Step 1: Investigate the nutrition status of all children aged 24 - 71 months in 10 preschools in 10 selected communes. Expecting 4500 targets in 10 examined preschools Step 2: After the investigative selection, participants that meet the standard will be invited to the study ( the communes selected can be narrowed if the target was hit). As soon as parents sign the consent paper, the study will move to the next step.
  Step 3: Groups will be divided to investigate activities. Creating a list for all participants that meet the criteria, with WHZ(Weight for Height Z-score)/BAZ(Body Mass Index for Age Z-score)<-0,5. Random selection based on age to ensure no significant difference in the nutritional index or related indicators in the group to assess the effectiveness of the intervention (divided by class/age). Then, randomly divided the participants by class into three large groups (300 targets per group)
Who Masked: Participant, Investigator
Masking Description: Control Group (300 participants): Children eat usual dietary(not using nutrient products) for 3 months. After that, they will use the product.
  Intervention Group (300 participants): Children eat usual dietary, but with 2 glasses of the nutrient product as the side meals. The product provides L-lysin, IgG 24h Colostrum, Calcium, Probiotics, HMO, DHA(Docosa Hexaenoic Acid), and Taurine within 3 months of use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Diet (No Intervention): (n=300): Children eat usual dietary (not using nutrient products) for 3 months. After that, they will use the products
- Colos Gain Dietary Supplement (Experimental): (n=300): Children eat usual dietary, but with 2 glasses of the nutrient product as the side meals. The product provides GOS(Galactooligosaccharides), Calcium, Probiotics, HMO, DHA, and Taurine within 3 months of use.
  Interventions: Dietary Supplement: Colos Gain

INTERVENTIONS:
Dietary Supplement: Colos Gain — Dietary Supplement: Colos Gain Colos Gain is a nutrient product made by VITADAIRY Dairy Joint Stock Company.
  Condition: Powder
  Color: White to light yellow
  Scent: The fresh scent of milk, gracious sugary smell.
  Date of use: 24 months from the manufactured date.
  Direction: Mix 5 spoons of Colos Gain (equal to 45 grams) with 180 ml of warm water (50˚C) which provides 210kcal (The energy density reaches 1kal/ml). Consume 2-3 glasses per day or follow the directions from the medical supervisors.
  The product should consume less than 1 hour. Do not let the child eat the leftovers of the previous meal.
  Preserve: Store in a clean, dry place, and keep away from direct sunlight. Opened can or package must be closed and used up within 3 weeks.
  Arms: Colos Gain Dietary Supplement

SUMMARY:
Evaluating the efficiency of using the nutrient production toward nutrition status (anthropometric index, the prevalence of wasting), digestive disorders, anorexia, and upper respiratory infections in children aged 24 - 71 months.

DETAILED DESCRIPTION:
The research involves a randomized controlled clinical trial (RCT), the plan is expected to conduct from 2022 to 2023 with over 600 children aged 24-71 months. The nutritional product produces a high amount of energy that provides over 468 kcal/100g; 12,5g/100g of protein; 12,5/100 of fat; 59,5g/100g of carbohydrate 1000ng/100g of IgG (immunoglobulin G) Colostrum; 15,3mg/100g of 2'FL HMO (health maintenance organization); 160mg/100g of MCT(Medium chain triglycerides) ; 3,7mg/100g of FOS(Fructo-Oligosaccharide) /Inulin; 810mg/100g of Lysine; 525mg/100g of Calcium; 55,6mg/100g of Magnesium; 5,6mg/100g of Iron; 3mg/100g of Zinc; 35,7µg/100g of Manganese; 8,1µg/100g of Selenium; 1290IU/100g of Vitamin A; 220 IU/100g of Vitamin D3; 33,1µg/100g of Vitamin K1; 510µg/100g of Vitamin B1; 700µg/100g of Vitamin B2; 360µg/100g of Vitamin B6; 1,4µg/100g Vitamin B12; 3120µg/100g of Acid Pantothenic; 62,7µg/100g of Acid Folic. 90 grams of the product which equals 2 packs (210ml x 2 per day) will supply about 33,0% - 43,6% of the required energy for children aged 2-5 years. Other 25 micronutrients and minerals include some essential vitamins such as Calcium 78,8 - 94,5 % RDAs, Iron 91-93% RDAs(recommended daily allowances), Vitamin A 86-103,2% RDAs, Zinc 56-66% RDAs, Vitamin D3 33% RDAs, Selenium 37-43% RDAs, Vitamin K1 43-50% RDAs, Folic Acid 38-56% RDAs. With other elements such as 2'FL HMO (15,3 mg), FOS/inulin (3700 mg), Choline ( 28 mg, Taurin 15,5 mg) ,colostrum IgG 24 1000mg. The study will be conducted at schools and homes: 600 children erratically divided into 2 groups, 1 group will use the product for 3 months (with the amount of use: twice per day, 45,0 grams each time). The product will be distributed to the students through the schools. Monitoring will be performed carefully by the commune and district Health Department and the Centers for Disease Control and Prevention weekly. The study aims to evaluate the efficiency of nutritional products toward nutrition status ( anthropometric index, the prevalence of wasting), digestive disorders, anorexia, and upper respiratory infections in children aged 24-71 months.

ELIGIBILITY:
Inclusion Criteria:

* Children between the age of 24 - 71 months old that currently study in 10 preschools in the area of 10 selected communes.
* The family volunteered for the child to participate in the study
* Currently residing at 10 selected communes (over 1 year of residing)
* Z-score WHZ/BAZ < - 0.5

Exclusion Criteria:

* Lactose intolerance
* Children with a history of allergies, congenital diseases
* Intellectual disability or are suffering from acute and chronic infectious diseases

Ages: 24 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Change of anthropometric indicators and nutrient status (wasting) | Up to 3 months of intervention
  Children in the intervention group will improve more with the anthropometric indicators (weight, height) than children in the control group.
  Weight is measured in kg with one decimal value by the Body composition analyzer called the TANITA scale. Children wear light clothes while measuring. A wooden stadiometer measures height by precisely 0.1cm.
  The nutrient status will be measure base on the changes in weight and height, also on
Change of digestive disorders, anorexia nervosa, and upper respiratory infections | From date of using the product until the date of first documented improvement, assessed up to 3 months
  Children in the intervention group improved more in digestive disorders, anorexia, and upper respiratory infections than in the control group.
  The changes in digestive disorders would illustrate in children defecating activities

SECONDARY OUTCOMES:
Body Mass Index, i.e. changes of Body Mass Index (BMI) | over 1 and 3 months
  Weight is measured in kg with one decimal value by the Body composition analyzer TANITA scale. The scale is checked and adjusted before use. Children wear light clothing, remove shoes and sandals, and sit or lie balanced, at the center of the scale. As soon as the balance is stable, read and write the result in kg and an odd number after the comma.
  A wooden stadiometer measures height by precisely 0.1cm. Children stand up straight, their eyes look straight, and the top of their head touches the wooden shelf fixed at a 0 cm position. The child's whole body ensures that 9 points touch the surface of the ruler: occipital, shoulder blade, buttocks, calf, and heel. The result is recorded in centimeters and an odd number after the comma.
  All data will be measured at the time T0 (at baseline) and T3 (after 3 months)
Change of weight for age Z-score | over 1 and 3 months
  Change of average weight for age Z Score and the difference between before intervention and after the intervention.
  Weight is measured in kg with one decimal value by the Body composition analyzer TANITA scale. The scale is checked and adjusted before use. Children wear light clothing, remove shoes and sandals, and sit or lie balanced, at the center of the scale. As soon as the balance is stable, read and write the result in kg and an odd number after the comma.
  Age of the child is calculated by subtracting the date of birth from the census date and classified according to WHO (World Health Organization) , 2006
Change of weight for height Z-score | over 1 and 3 months
  Change of average weight for height Z Score and the difference between before intervention and after the intervention.
  Weight is measured in kg with one decimal value by the Body composition analyzer TANITA scale. The scale is checked and adjusted before use. Children wear light clothing, remove shoes and sandals, and sit or lie balanced, at the center of the scale. As soon as the balance is stable, read and write the result in kg and an odd number after the comma.
  A wooden stadiometer measures height by precisely 0.1cm. Children stand up straight, their eyes look straight, and the top of their head touches the wooden shelf fixed at a 0 cm position. The child's whole body ensures that 9 points touch the surface of the ruler: occipital, shoulder blade, buttocks, calf, and heel. The result is recorded in centimeter and an odd number after the comma.
Change of height for age Z-score | over 1 and 3 months
  Change of average height for age Z Score and the difference between before intervention and after the intervention.
  A wooden stadiometer measures height by precisely 0.1cm. Children stand up straight, their eyes look straight, and the top of their head touches the wooden shelf fixed at a 0 cm position. The child's whole body ensures that 9 points touch the surface of the ruler: occipital, shoulder blade, buttocks, calf, and heel. The result is recorded in centimeters and an odd number after the comma.
  Age of the child is calculated by subtracting the date of birth from the census date, and classified according to WHO, 2006
Changes in the percentage of children have anorexia, upper respiratory infections or gastrointestinal diseases | over 1 and 3 months
  Changes in the percentage of anorexia, the percentage of gastrointestinal diseases (diarrhea, constipation), and anorexia above after intervention. The changes in digestive disorders would demonstrate in children defecating activities

OTHER OUTCOMES:
Changes in the percentage of wasted and malnutrition children | over 1 and 3 months
  Changes in the risk of wasting and malnutrition after 1, 2, and 3 months of intervention. Data were entered using Epidata 3.1 software. Data analysis using the software called SPSS 18.0. Anthropometric data were processed using Anthro software from WHO, 2006. Statistics were used to analyze the data of the squared test (χ2-test) and Fisher's exact test to compare the difference between the samples. ratio; Mc Nemar -test compares the difference in the percentage of malnutrition of each study group before and after the intervention. The rate of children got wasting and malnutrition will decrease as the body index increase over time. The measurement would be done by a TANITA scale and a wooden stadiometer.

CONTACTS AND LOCATIONS:
Overall Officials: Division of Planning National Institute of Nutrition, Principal Investigator — National Institute of Nutrition, Vietnam
Locations (1):
- Yen Bai Province Obstetrics and Children's Hospital, Yên Bái, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about the organization in which this study is conducted. The Division of Planning is responsible to plan and implement the project. — http://viendinhduong.vn/en/home.html